CLINICAL TRIAL: NCT01727336
Title: A Phase 2 Randomized, Double-Blind Study of Dalantercept and Axitinib Compared to Placebo and Axitinib in Patients With Advanced Renal Cell Carcinoma
Brief Title: Study of Dalantercept and Axitinib in Patients With Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the sponsor following unblinding of the Progression Free Survival endpoint.
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A041-04; ACE-041 (Other: Acceleron Pharma Inc.)
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2021-09

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — ALK1-Fc fusion protein, human; Axitinib

STUDY DESIGN:
Intervention Model Description: Part 1 of the study involved a dose escalation phase to select a dose for Part 2 of the study. In Part 1, a total of 29 subjects escalated through 3 dose levels of dalantercept: 0.6, 0.9 and 1.2 mg/kg once every 3 weeks. In Part 2, dalantercept (0.9 mg/kg once every 3 weeks) plus axitinib 5 mg PO BID) was compared with placebo plus axitinib 5 mg PO BID. Part 2 enrolled 131 subjects for a total of 160 subjects in the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dalantercept 0.9 mg/kg plus axitinib (Experimental): Subcutaneous (SC) injection of dalantercept 0.9 mg/kg once every 3 weeks and oral axitinib 5 mg BID for continuous dosing.
  Interventions: Drug: Dalantercept and axitinib
- Placebo plus axitinib (Placebo Comparator): Subcutaneous injection of normal saline once every 3 weeks and oral axitinib 5 mg BID for continuous dosing
  Interventions: Drug: Placebo and axitinib
- Dalantercept 0.6 mg/kg (Experimental): Part 1 dose escalation arm 0.6 mg/kg dalantercept once every 3 weeks
  Interventions: Drug: Dalantercept and axitinib
- Dalantercept 0.9 mg/kg (Experimental): Part 1 dose escalation arm 0.9 mg/kg dalantercept once every 3 weeks
  Interventions: Drug: Dalantercept and axitinib
- Dalantercept 1.2 mg/kg (Experimental): Part 1 dose escalation arm 1.2 mg/kg dalantercept once every 3 weeks
  Interventions: Drug: Dalantercept and axitinib
- Dalantercept 1.5 mg/kg (Experimental): Part 1 dose escalation arm 1.5 mg/kg dalantercept once every 3 weeks
  Interventions: Drug: Dalantercept and axitinib

INTERVENTIONS:
Drug: Dalantercept and axitinib
  Other Names: ACE-041, Inlyta
  Arms: Dalantercept 0.6 mg/kg; Dalantercept 0.9 mg/kg; Dalantercept 0.9 mg/kg plus axitinib; Dalantercept 1.2 mg/kg; Dalantercept 1.5 mg/kg
Drug: Placebo and axitinib
  Other Names: Inlyta
  Arms: Placebo plus axitinib

SUMMARY:
The purpose of Part 1 of this study is to evaluate the safety and tolerability of dalantercept in combination with axitinib in patients with advanced renal cell carcinoma (RCC) to determine the recommended dose level of dalantercept in combination with axitinib for Part 2.

The purpose of Part 2 of this study is to determine whether treatment with dalantercept in combination with axitinib prolongs progression free survival (PFS) compared to axitinib alone in patients with advanced renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
In Part 1 of the study, groups of subjects received escalating doses of dalantercept; 0.6, 0.9 and 1.2 mg/kg in sequential groups. All subjects received concurrent axitinib 5 mg PO BID. A total of 29 subjects were enrolled i Part 1 of the study.

In Part 2, dalantercept at 0.9 mg/kg once every 3 weeks plus axitinib 5 mg PO BID was compared to placebo plus axitinib 5 mg PO BID. A total of 131 subjects were enrolled in Part 2 for a total of 160 in the study

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed, advanced, predominantly clear cell renal cell carcinoma (RCC).
* Part 1: Progression of disease following up to three lines of prior therapy, including at least one approved VEGF receptor tyrosine kinase inhibitor for RCC. Adjuvant therapy is permitted as one line of prior therapy.
* Part 2: Progression of disease following one VEGF pathway inhibitor for RCC (e.g. sunitinib, pazopanib, sorafenib, bevacizumab, tivozanib, or cabozantinib) inclusive of adjuvant therapy if there was documented disease progression during treatment. Patients may have received one additional line of an approved mTOR kinase inhibitor (e.g. everolimus, temsirolimus). Prior exposure to investigational and/or approved anticancer immune therapies is permitted.
* A minimum of 1 week since the last dose of prior therapy (a minimum of 4 weeks since anticancer immune therapy or bevacizumab +/- interferon).
* Measurable disease that is evaluable by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Clinical laboratory values within acceptable ranges within 72 hours prior to study day 1.

Key Exclusion Criteria:

* Clinically significant organ/system disease unrelated to RCC that in the judgment of the investigator should preclude treatment with dalantercept or axitinib.
* Clinically significant cardiovascular risk.
* Known CNS metastases or leptomeningeal disease:

For Part 1, patients with CNS metastases treated with whole brain radiotherapy, gamma knife, and/or surgery who are considered stable by CNS imaging and are not being treated with corticosteroids 6 weeks prior to study day 1 may be enrolled.

For Part 2, patients with CNS metastases treated stereotactic radio-surgery (SRS), and/or surgery who are considered stable by CNS imaging for at least 2 months prior to enrollment and are not being treated with corticosteroids 6 weeks prior to study day 1 may be enrolled.

* Any active malignancy, other than RCC, for which chemotherapy or other anti-cancer therapy is indicated. Patients with adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 3 years will be permitted.
* Any lesion invading or having encasement ≥ 180 degrees around the wall of a major blood vessel as assessed by computed tomography (CT) scan and/or magnetic resonance imaging (MRI).
* Radiotherapy within 2 weeks prior to study day 1.
* Lack of recovery from toxic effects of previous treatment for RCC ≤ grade 1 with the exception of alopecia, unless stabilized under adequate medical control.
* Patients undergoing renal dialysis.
* Major surgery within 4 weeks prior to study day 1 (patients must have recovered completely from any previous surgery prior to study day 1).
* Any active infection requiring antibiotic therapy within 2 weeks of study day 1.
* Anti-coagulation therapy. Aspirin, other anti-platelet agents, and low molecular weight heparin are permitted unless the investigator deems the patient is at a significant risk for bleeding.
* Current use or anticipated inability to avoid potent CYP3A4/5 inhibitors or inducers (please refer to the Inlyta® [axitinib] prescribing information) during participation in the study.
* Peripheral edema requiring medical intervention within 2 weeks prior to study day 1.
* Bleeding diathesis including clinically significant platelet disorders or active hemoptysis (defined as bright red blood of ≥ 1/2 teaspoon [2.5 mL] in any 24 hour period) within 6 months prior to study day 1. For clinically significant epistaxis within 4 weeks prior to study day 1, no risk of further bleeding must be clearly documented.
* Known history of hereditary hemorrhagic telangiectasia (HHT).
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections or positive human immunodeficiency virus (HIV) antibody results. Patients with sustained virologic response to HCV treatment or immunity to HBV from prior infection without cirrhosis may be included.
* History of severe (defined as ≥ grade 3, using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 4.0 [NCI-CTCAE] v4 current active minor version) allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients (10 mM Tris buffered saline) in the investigational agent.
* Any prior treatment with dalantercept or any other agent targeting ALK1 pathway.
* Any prior treatment with axitinib.
* A morbidity (per the prescribing information) that would require starting a patient at a reduced dose of axitinib.
* Treatment with another investigational drug (with the exception of anticancer immune therapy) or device, or approved therapy for investigational use, within 5 times the half-life of the drug or within 3 weeks prior to study day 1 if the half life is not known.
* Pregnant or lactating female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - University of California Irvine Medical Center, Irvine, California
  - University of California, Los Angeles (UCLA) - Institute of Urologic Oncology, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Loyola University Chicago, Chicago, Illinois
  - Indiana University Health Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Cancer Center Hackensack UMC, Hackensack, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - North Shore LIJ Center for Advance Medicine, Lake Success, New York
  - Mem Sloan Kettering Cancer Center, New York, New York
  - NYU Cancer Institute, New York, New York
  - Levin Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Saint Luke's University Health Network, Bethlehem, Pennsylvania
  - Penn State Milton S- Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology-South Austin, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology - Tyler and Longview, Tyler, Texas
  - Shenandoah Oncology P.C., Winchester, Virginia
  - University of Wisconsin, Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- [Derived] Voss MH, Bhatt RS, Vogelzang NJ, Fishman M, Alter RS, Rini BI, Beck JT, Joshi M, Hauke R, Atkins MB, Burgess E, Logan TF, Shaffer D, Parikh R, Moazzam N, Zhang X, Glasser C, Sherman ML, Plimack ER. A phase 2, randomized trial evaluating the combination of dalantercept plus axitinib in patients with advanced clear cell renal cell carcinoma. Cancer. 2019 Jul 15;125(14):2400-2408. doi: 10.1002/cncr.32061. Epub 2019 Apr 5. PMID 30951193

FDAAA 801 VIOLATIONS:
- Correction Confirmed — The responsible party has corrected the violation. — issued 2021-12-13, released 2021-09-14, posted 2021-12-14
- Violation Identified — Failure to Submit. The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2021-04-27, released 2019-01-09, posted 2021-04-29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Part 1 dose escalation portion of the study, 4 dose levels of dalantercept plus an expansion cohort were planned. However, dose escalation was suspended following the 1.2 mg/kg dose level and additional subjects were added to the 1.2 mg/kg dose cohort, which represented the expansion; no subjects were enrolled in the 1.5 mg/kg dose level.
Groups:
- Part 1 Dalantercept 0.6 mg/kg: Dose escalation cohort 1: dalantercept 0.6 mg/kg plus axitinib 5 mg PO BID
- Part 1 Dalantercept 0.9 mg/kg: Dose escalation cohort 2: dalantercept 0.9 mg/kg plus axitinib 5 mg PO BID
- Part 1: Dalantercept 1.2 mg/kg: Part 1 cohort 3: dalantercept 1.2 mg/kg plus axitinib 5 mg PO BID
- Part 1: Dalantercept 1.5 mg/kg: Dose escalation cohort 4: dalantercept 1.5 mg/kg
- Part 2: Dalantercept 0.9 mg/kg Plus Axitinib: Subcutaneous (SC) injection of Dalantercept once every 3 weeks and oral axitinib 5 mg PO BID for continuous dosing.
- Part 2: Placebo Plus Axitinib: Subcutaneous injection of normal saline once every 3 weeks and oral axitinib 5 mg PO BID for continuous dosing
Period: Part 1 Dalantercept Dose Escalation
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg | Part 1: Dalantercept 1.5 mg/kg | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Started | 6 | 9 | 14 | 0 | 0 | 0
Completed | 3 | 7 | 6 | 0 | 0 | 0
Not Completed | 3 | 2 | 8 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 3 | 0 | 0 | 0
Period: Part 2 Blinded
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg | Part 1: Dalantercept 1.5 mg/kg | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Started | 0 | 0 | 0 | 0 | 63 | 68
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 63 | 68
Not completed — Death | 0 | 0 | 0 | 0 | 20 | 16
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 42 | 44
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 4
Not completed — use of prohibited medications | 0 | 0 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled into the 1.5 mg/kg dose escalation cohort
Groups:
- Part 1 Dalantercept 0.6 mg/kg: Dose escalation cohort 1: dalantercept 0.6 mg/kg
- Part 1 Dalantercept 0.9 mg/kg: Dose escalation cohort 2: dalantercept 0.9 mg/kg
- Part 1 Dalantercept 1.2 mg/kg: Dose escalation cohort 3: dalantercept 1.2 mg/kg
- Part 1 Dalantercept 1.5 mg/kg: Dose escalation cohort 4: dalantercept 1.5 mg/kg
- Part 2 Dalantercept 0.9 mg/kg Plus Axitinib: Subcutaneous (SC) injection of Dalantercept once every 3 weeks and oral axitinib 5 mg BID for continuous dosing.
- Total: Total of all reporting groups
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1 Dalantercept 1.2 mg/kg | Part 1 Dalantercept 1.5 mg/kg | Part 2 Dalantercept 0.9 mg/kg Plus Axitinib | Placebo Plus Axitinib | Total
Number analyzed (Participants) | 6 | 9 | 14 | 0 | 63 | 68 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (7.2) | 56.2 (9.2) | 61.5 (10.9) |  | 62.8 (8.1) | 58.9 (10.1) | 60.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 |  | 22 | 28 | 56
  Male | 5 | 7 | 11 |  | 41 | 40 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 |  | 1 | 6 | 9
  Not Hispanic or Latino | 6 | 8 | 13 |  | 58 | 58 | 143
  Unknown or Not Reported | 0 | 0 | 0 |  | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 14 |  | 63 | 68 | 160

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events as a Measure of Safety and Tolerability.
Description: Outcome measure is intended for Part 1 of the study in order to determine recommended dose level for Part 2.
Time Frame: Assessed from time of first dose to approximately 30 days after last dose. Participants were allowed to remain on treatment until documented disease progression. The time frame for Part 1 of the study was up to 21.6 months
Population: Safety Analysis Set (SAF) consisted of all patients who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Dalantercept 0.6 mg/kg: Part 1 cohort 1; dalantercept 0.6 mg/kg plus axitinib 5 mg PO BID
- Part 1 Dalantercept 0.9 mg/kg: Part 1 cohort 2; dalantercept 0.9 mg/kg plus axitinib 5 mg PO BID
- Part 1 Dalantercept 1.2 mg/kg: Part 1 cohort 3; dalantercept 1.2 mg/kg plus axitinib 5 mg PO BID
- Part 1 Dalantercept 1.5 mg/kg: Part 1 cohort 1; dalantercept 1.5 mg/kg plus axitinib 5 mg PO BID
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1 Dalantercept 1.2 mg/kg | Part 1 Dalantercept 1.5 mg/kg
Number analyzed (Participants) | 6 | 9 | 14 | 0
Participants | 6 | 9 | 14 |
Statistical Analysis 1: Comparison: Part 1 Dalantercept 0.6 mg/kg vs Part 1 Dalantercept 0.9 mg/kg vs Part 1 Dalantercept 1.2 mg/kg vs Part 1 Dalantercept 1.5 mg/kg; Test type: Other; recommended dose for Part 2 = 0.9 — The recommended dose level for Part 2 was determined to be 0.9 mg/kg

2. Primary Outcome: Part 2: Progression Free Survival (PFS).
Description: PFS was defined as the time from randomization to the date of first documentation of disease progression based on RECIST (version 1.1) or to death due to any cause, whichever occurred first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
  RECIST 1.1 defines disease progression as an increase of at least a 20% in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression)
Time Frame: Progression free survival is defined as the time from the date of the randomization to the first documented disease progression (according to RECIST v1.1) or death due to any cause. The Time frame for Part 2 was up to 29.0 months
Population: The All Treated Set (ATS) included all randomized patients who received any study drug
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 2: Dalantercept 0.9 mg/kg Plus Axitinib: Subcutaneous (SC) injection of Dalantercept 0.9 mg/kg once every 3 weeks and Oral axitinib 5 mg BID for continuous dosing.
- Part 2: Placebo Plus Axitinib: Subcutaneous injection of normal saline once every 3 weeks and oral axitinib 5 mg BID for continuous dosing
Arm/Group | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 58 | 61
Months | 6.8 [4.5 to 9.4] | 5.6 [3.3 to 8.3]

3. Secondary Outcome: Part 1: Progression Free Survival (PFS).
Description: PFS was defined as the time from randomization to the date of first documentation of disease progression based on RECIST (version 1.1) or to death due to any cause, whichever occurred first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: The time frame for Part 1 of the study was up to 21.6 months
Population: Full Analysis Set; all subjects randomized in Part 1 of the study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 6 | 9 | 14
Months | 5.5 [1.3 to 20.6] | 21.6 [2.8 to 21.6] | 6.9 [2.7 to 20.7]

4. Secondary Outcome: Part 1: Overall Survival (OS). [The Time Frame for Part 1 of the Study Was up to 21.6 Months]
Description: Percentage of Part 1 subjects alive at the end of Part 1 of the study. [The time frame for Part 1 of the study was up to 21.6 months]
Time Frame: Up to 21.6 months
Population: Full Analysis Set; all subjects randomized in Part 1 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 6 | 9 | 14
Participants | 4 | 7 | 9

5. Secondary Outcome: Part 1: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the number and percentage of patients who have a partial response (PR) or complete response (CR) to therapy. A CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. A PR is defined as a decrease of at least a 30% in the sum of diameters of target lesions, taking as reference the baseline sum diameters. As no subjects in Part 1 experienced a CR, the ORR in Part 1 is defined by the PR
Time Frame: Up to 21.6 months from randomization in Part 1 of the study
Population: Full Analysis Set; all subjects randomized in Part 1 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 6 | 9 | 14
Participants | 2 | 3 | 2

6. Secondary Outcome: Part 1: Disease Control Rate (DCR)
Description: The number and percentage of patients whose disease shrinks or remains stable. DCR is the sum of the complete, partial and stable disease rates.
Time Frame: From randomization up to 21.6 months in Part 1 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 6 | 9 | 14
Participants | 3 | 5 | 6

7. Secondary Outcome: Part 1: Duration of Response (DoR)
Description: Response duration is measured from the time measurement criteria are first met for objective response until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study.
Time Frame: From randomization up to 21.6 months in Part 1 of the study.
Population: Full Analysis Set; all subjects randomized in Part 1 of the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Dalantercept 0.6 mg/kg | Part 1 Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg
Number analyzed (Participants) | 6 | 9 | 14
months | 3 [2.8 to 21.6] | 6.9 [6.9 to 21.6] | 10 [8.8 to 11.1]

8. Secondary Outcome: Part 2: Progression Free Survival (PFS) for the Subset of Participants With 2 or More Lines of Prior Systemic Chemotherapy
Description: Progression Free Survival (PFS) for the subset of participants with 2 or more lines of prior systemic chemotherapy. PFS was based upon RECIST 1.1 assessment, as described in outcome measure 2.
Time Frame: as for outcome 2
Population: Subgroup of Part 2 participants:
  24 of 63 participants in the dalantercept arm and 22 of 68 participants in the placebo arm had at least 2 lines of prior systemic chemotherapy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 24 | 22
Months | 8.1 [3.6 to 10.5] | 7.0 [2.8 to 9.5]

9. Secondary Outcome: Part 2: Overall Survival.
Description: The number of months from the date of randomization to the date of death.
Time Frame: Patients to be contacted every 3 months for up to 12 months (anticipated) for survival follow-up, as well as tumor assessment scans if progression of disease has not previously been documented. The time frame for Part 2 was up to 29.0 months
Population: The All Treated Set (ATS) included all randomized patients who received any study drug
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 58 | 61
Months | 13.0 [9.3 to 14.5] | 14.7 [7.3 to 20.0]

10. Secondary Outcome: Part 2: Objective Response Rate.
Description: Objective response rate (ORR) is defined as the number and percentage of patients who have a partial response (PR) or complete response (CR) to therapy. A CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. A PR is defined as a decrease of at least a 30% in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessed at 30 days after last dose of study drug; up to 29.0 months for Part 2 of the study
Population: The All Treated Set (ATS) included all randomized patients who received any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 58 | 61
Participants | 11 | 15

11. Secondary Outcome: Part 2: Duration of Response
Description: as for outcome 7
Time Frame: Assessed at 30 days after the last dose of study drug; up to 29.0 months for Part 2 of the study.
Population: The All Treatment Set (ATS) included all randomized patients who received any study drug. Please see Outcome Measure 5 for Objective Response Rate data. Since there were too few participants with events, an estimation of response duration was not able to be calculated due to the early termination of the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 58 | 61
Months | NA [NA to NA] — too few participants with events were available for an estimation of response duration due to the early termination of the study | NA [NA to NA] — too few participants with events were available for an estimation of response duration due to the early termination of the study

12. Secondary Outcome: Part 2: Disease Control Rate.
Description: as for outcome 6
Time Frame: Assessed at 30 days after last dose of study drug. The time frame for Part 2 was up to 29.0 months
Population: The All Treated Set (ATS) included all randomized patients who received any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 58 | 61
Participants | 48 | 50

13. Other Pre Specified Outcome: Part 1: Exploratory PD - Serum BMP9
Description: Exploratory analysis. Absolute change from baseline in serum Bone Morphogenetic Protein 9 (BMP9)
Time Frame: From randomization up to 21.6 months in Part 1 of the study
Population: All subjects randomized to Part 1 of the study and treated with at least 1 dose of dalantercept. Given the high degree of variability in serum BMP9 levels in study subjects [Baseline value 23.55 ng/mL (SD 20.54 ng/mL)] and the relative small numbers of subjects in each treatment arm, it was decided that the best way to understand a treatment effect was to conduct a pooled analysis of all 29 Part 1 subjects for the comparison of change from Baseline.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1 Participants: Pooled number of Part 1 participants across the dose escalation groups 0.6 mg/kg (N=6), 0.9 mg/kg (N=9) and 1.2 mg/kg (N=14); total N=29 subjects
Arm/Group | Part 1 Participants
Number analyzed (Participants) | 29
ng/mL | -11.5 (2.58)

14. Other Pre Specified Outcome: Part 2: PD Biomarker Activities.
Description: Exploratory analysis. Absolute change from baseline in serum Bone Morphogenetic Protein 9 (BMP9)
Time Frame: Assessed at 30 days after the last dose of dalantercept ± 10 days. The time frame for Part 2 was up to 29.0 months.
Population: The All Treated Set (ATS) included all randomized patients who received any study drug, and for whom sufficient blood sample was available to assess the exploratory biomarker.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
Number analyzed (Participants) | 45 | 46
pg/mL | -53.34 (37.87) | 8.55 (86.32)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the initial study drug administration on Cycle 1, Day 1 (C1D1) until 30 days after the last study drug administration for each subject on study, up to a total of 29.0 months of study drug exposure
Description: Analyses of adverse events were carried out on the Safety Analysis Set, defined as all participants who received at least one dose of study drug.
  There were no subjects enrolled in Part 1 cohort 4 (1.5 mg/kg dalantercept), thus no subjects were at risk for adverse events
Groups:
- Part 1: Dalantercept 0.6 mg/kg: Part 1 cohort 1: dalantercept 0.6 mg/kg plus axitinib 5 mg PO BID
- Part 1: Dalantercept 0.9 mg/kg: Part 1 cohort 1: dalantercept 0.9 mg/kg plus axitinib 5 mg PO BID
- Part 1: Dalantercept 1.2 mg/kg: Part 1 cohort 1: dalantercept 1.2 mg/kg plus axitinib 5 mg PO BID
- Part 1: Dalantercept 1.5 mg/kg: Part 1 cohort 1: dalantercept 1.5 mg/kg plus axitinib 5 mg PO BID
Arm/Group | Part 1: Dalantercept 0.6 mg/kg | Part 1: Dalantercept 0.9 mg/kg | Part 1: Dalantercept 1.2 mg/kg | Part 1: Dalantercept 1.5 mg/kg | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib | Part 2: Placebo Plus Axitinib
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/9 | 5/14 | 0/0 | 20/63 | 16/68
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/9 | 6/14 | 0/0 | 19/62 | 16/64
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 14/14 | 0/0 | 61/62 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1: Dalantercept 0.6 mg/kg (N=6) | Part 1: Dalantercept 0.9 mg/kg (N=9) | Part 1: Dalantercept 1.2 mg/kg (N=14) | Part 1: Dalantercept 1.5 mg/kg (N=0) | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib (N=62) | Part 2: Placebo Plus Axitinib (N=64)
pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
PLeural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Periportal oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0/58 | 0/61
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bile duct stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gate disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Transaminase increase (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dalantercept 0.6 mg/kg (N=6) | Part 1: Dalantercept 0.9 mg/kg (N=9) | Part 1: Dalantercept 1.2 mg/kg (N=14) | Part 1: Dalantercept 1.5 mg/kg (N=0) | Part 2: Dalantercept 0.9 mg/kg Plus Axitinib (N=62) | Part 2: Placebo Plus Axitinib (N=64)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 0 (0) | 54 (54) | 55 (55)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 0 | 38 (38) | 40 (40)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 | 0 | 24 (24) | 28 (28)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 18 (18) | 18 (18)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 3 (3) | 0 | 13 (13) | 16 (16)
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 8 (8) | 15 (15)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 (6) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1) | 3 (3) | 0 | 4 (4) | 5 (5)
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7 (7) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 (2) | 5 (5)
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 (3) | 4 (4)
Fatigue (General disorders) | 4 (4) | 5 (5) | 10 (10) | NA | 35 (35) | 47 (47)
Chills (General disorders) | 0 | 0 | 0 | 0 | 8 (8) | 5 (5)
Oedema peripheral (General disorders) | 0 | 3 (3) | 6 (6) | 0 | 24 (24) | 14 (14)
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 6 (6) | 6 (6)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 7 (7) | 5 (5)
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 7 (7) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 | 11 (11) | 25 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 | 24 (24) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 16 (16) | 13 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 7 (7) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 6 (6) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 3 (3) | 0 | 6 (6) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 (2) | 3 (3) | NA | 17 (17) | 19 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 10 (10) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 14 (14) | 9 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 | 7 (7) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 9 (9) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 (4) | 6 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 (3) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 (3) | 7 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 (2) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 (4) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 3 (3) | 0 | 15 (15) | 15 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 (4) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 (2) | 1 (1) | 0 | 6 (6) | 8 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 6 (6) | 6 (6)
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 (5) | 6 (6)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 5 (5) | 1 (1) | 0 | 6 (6) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 (2) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 6 (6)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0 | 13 (13) | 20 (20)
Blood creatinine increased (Investigations) | 0 | 0 | 6 (6) | 0 | 21 (21) | 11 (11)
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 5 (5) | 7 (7)
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 7 (7) | 5 (5)
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 2 (2) | 9 (9)
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 5 (5) | 5 (5)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 (2) | 5 (5)
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 6 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 5 (5) | 0 | 23 (23) | 20 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 5 (5) | 13 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 7 (7) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6 (6) | 8 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 2 (2) | 0 | 7 (7) | 6 (6)
Headache (Nervous system disorders) | 0 | 1 (1) | 2 (2) | 0 | 14 (14) | 21 (21)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 7 (7) | 6 (6)
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 (4) | 6 (6)
Hypertension (Vascular disorders) | 0 | 2 (2) | 1 (1) | 0 | 13 (13) | 30 (30)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 (2) | 6 (6)
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 (3) | 4 (4)
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 4 (4) | 11 (11)
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 9 (9) | 2 (2)
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 (4) | 9 (9)
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 6 (6) | 5 (5)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 (2) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 3 (3) | 0 | 13 (13) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 (1) | 3 (3) | 0 | 4 (4) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 | 2 (2) | 3 (3) | 0 | 8 (8) | 12 (12)
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 2 (2) | 7 (7)

LIMITATIONS AND CAVEATS:
All 131 patients in Part 2 discontinued from the study; the most frequent reasons were (i) study terminated at the discretion of the sponsor [86 patients (65.6%)] and (ii) death [36 patients (27.5%)]. The discontinuations prior to planned sample collections, as outlined in the protocol schedule of events, precluded the ability to carry out all planned analyses, including but not limited to PK analyses. Dalantercept PK in patients with advanced cancer has been reported previously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT01727336/Prot_SAP_000.pdf